CLINICAL TRIAL: NCT00893295
Title: Increasing Colon Cancer Screening in Primary Care Among African Americans
Brief Title: Increasing Colorectal Cancer Screening in African Americans
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Ronald Myers, Jefferson Medical College of Thomas Jefferson University
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Screening
Other Study IDs: CDR0000635953; TJUH-RSGT-08-017-01-CPPB; 08G.89
Record Dates: First submitted 2009-05-02; First posted 2009-05-05 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Barium Enema; Sigmoidoscopy

INTERVENTIONS:
Other: informational intervention
Other: medical chart review
Other: screening questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: barium enema injection
Procedure: colon imaging study
Procedure: screening colonoscopy
Procedure: sigmoidoscopy

SUMMARY:
RATIONALE: Screening may help doctors find colorectal cancer sooner, when it may be easier to treat. Finding out what affects a patient's decision to undergo screening tests may help increase the number of patients who undergo regular screening for cancer. It is not yet known whether personalized invitations to undergo colorectal cancer screening are more effective than standard screening reminders.

PURPOSE: This randomized phase III trial is studying ways to increase colorectal cancer screening in African Americans.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the intervention impact on colorectal cancer (CRC) screening utilization over a 6-month observation period in African-American participants.
* To assess the intervention impact on CRC screening preference, classified into three levels (i.e., "decided not to screen or never heard of," "undecided," or "decided to screen"), based on data obtained from both the endpoint chart audit and the endpoint survey.
* To assess intervention impact on population health-management representations related to CRC screening, as assessed by perceived salience and coherence and self-efficacy related to CRC screening measured with 6 to 10 Likert-type items on both the baseline and endpoint surveys.
* To analyze intervention cost-effectiveness, from the societal perspective and from the more limited perspective of the provider and payer, focusing on the average and incremental cost per additional person who is compliant (i.e., has a CRC screening test during the observation period) for each alternative intervention and estimate the cost per life-year saved.

OUTLINE: This is a multicenter study. Participants are stratified according to practice. Participants are randomized to 1 of 2 intervention arms.

* Arm I (standard-intervention group): Participants receive a personalized screening invitation letter encouraging selection and performance of one of the screening tests, a generic colorectal cancer (CRC) screening informational booklet, stool blood testing (SBT) cards, and instructions for arranging a colonoscopy screening appointment. After 45 days, participants who have not been screened receive a reminder letter.
* Arm II (tailored-navigation intervention group): Participants receive a CRC screening invitation letter and materials that are tailored to the individual's preferred screening test strategy (i.e., SBT; SBT and instructions for arranging flexible sigmoidoscopy, instructions for arranging flexible sigmoidoscopy; or instructions for arranging colonoscopy). After 30 days, participants who have not been screened will receive a reminder by telephone. Those participants who have undergone screening will be congratulated for taking the time and preventative action, and be encouraged to continue future screenings. After 45 days, participants who have not been screened receive a reminder letter.

Participants are assessed by a baseline survey consisting of personal background, cognitive and psychological representations, social support and influence, intention, and decision stage related to screening SBT and colonoscopy preference. Data obtained from the endpoint survey assessing whether participants and their providers discussed CRC screening before the study and opinions about the intervention, and an endpoint chart audit to gather data on participant CRC screening exam dates and exam results (i.e., screening SBT, flexible sigmoidoscopy, colonoscopy, double-contrast barium enema [DCBE] x-ray) are assessed for group differences.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* African-American participants who receive medical care in a large, urban primary care practice setting and are eligible for colorectal cancer (CRC) screening
* Noncompliant with CRC screening in terms of American Cancer Society guidelines
* Attended an office visit within the past 2 years

PATIENT CHARACTERISTICS:

* No family history of colorectal cancer diagnosed before the age of 60 years
* No prior diagnosis of colorectal neoplasia (cancer or polyps) or inflammatory bowel disease

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 896 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Intervention impact on colorectal cancer (CRC) screening utilization over the 6-month observation period

SECONDARY OUTCOMES:
Intervention impact on CRC screening preference, based on data obtained from both the endpoint chart audit and the endpoint survey
Intervention impact on population health-management representations related to CRC screening, as assessed by perceived salience and coherence and self-efficacy-related CRC screening measured with 6 to 10 Likert-type items on both the baseline and end ...

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Myers, PhD, Principal Investigator — Jefferson Medical College of Thomas Jefferson University
Locations (1):
- Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania, United States